CLINICAL TRIAL: NCT03618316
Title: An Open-label, One-sequence Study to Assess the Effect of Repeated Oral Doses of Cimetidine on the Single Dose Pharmacokinetics, Safety and Tolerability of Imeglimin in Healthy Caucasian Subjects
Brief Title: Effect of Cimetidine on the PK of Imeglimin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PXL008-023
Record Dates: First submitted 2018-06-08; First posted 2018-08-07 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: pharmacokinetics; Drug-drug interaction
MeSH Terms: interventions — imeglimin; Cimetidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label imeglimin + cimetidine (Experimental): Day 1: single oral dose of 1,500 mg imeglimin Day 5 to Day 10 inclusive: repeated doses of 400 mg cimetidine twice daily Day 8: second 1,500 mg dose of imeglimin together with the morning dose of cimetidine
  Interventions: Drug: Imeglimin; Drug: Cimetidine

INTERVENTIONS:
Drug: Imeglimin — 2 singles oral doses of imeglimin 1,500 mg (one at day 1 and one at day 8)
Drug: Cimetidine — 400 mg of cimetidine bid from Day 5 to Day 10

SUMMARY:
The trial is an open-label assessment of the interaction of imeglimin with cimetidine. Up to 16 healthy men and women will receive a single oral dose of 1,500 mg imeglimin alone followed by a second dose of imeglimin during repeated doses of 400 mg cimetidine taken twice daily for 6 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI : 18.5-29.9
* Body weight ≥ 60 kg
* willing to use reliable contraception
* able to give fully informed written consent.

Exclusion Criteria:

* Pregnant or lactating woman, or sexually active woman of child-bearing potential not using reliable contraception
* Clinically relevant abnormal findings at the screening assessment
* Clinically significant vital signs outside the acceptable range at screening
* Clinically relevant abnormal medical history, surgery or concurrent medical condition
* Acute or chronic illness
* Estimated glomerular filtration rate less than 80 mL/min/1.73 m2
* Severe adverse reaction to any drug or sensitivity to the trial medication or its components
* Significant food allergy; vegetarian or vegan
* Participation in other clinical trials of unlicensed or prescription medicines, or loss of more than 400 mL blood, within the 3 months before first dose of trial medication
* Drug or alcohol abuse
* Smoking of more than 5 cigarettes daily
* Possibility that subject will not cooperate
* Positive test for hepatitis B & C, HIV
* Objection by a General Practitioner

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Caucasian
Enrollment: 16 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
PK parameters of imeglimin | At Day 1
  Cmax: peak plasma concentration after dosing

SECONDARY OUTCOMES:
PK parameters of imeglimin | From day 1 to day 3
  AUC last:area under the concentration-time curve
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | from day 1 to day 17
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom